CLINICAL TRIAL: NCT04545125
Title: Optimising the Care and Treatment Pathways for Older Patients Facing Major Gastrointestinal Surgery.
Acronym: OCTAGON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: STH20694
Record Dates: First submitted 2020-08-24; First posted 2020-09-10 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-09

CONDITIONS: Old Age; Debility; Gastro-Intestinal Disorder
MeSH Terms: conditions — Frailty; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The UK population is ageing. Whilst many people remain active and in good health as they get older, getting older is associated with the onset of many common medical conditions, as well as memory and mobility problems. There is a natural decline in heart and lung fitness with age, although this may be slowed by regular exercise and physical activity. The majority of digestive system problems that require operations (such as bowel cancer) are more common in older people. These operations can reduce an older person's ability to look after themselves and their quality of life. In some cases there is a trade-off between major surgery and a smaller operation or procedure with a lower chance of cure, but a faster rate of recovery and fewer problems immediately after the procedure. (Examples of smaller operations include bringing the bowel out onto the abdominal wall; creating a 'stoma'. Examples of procedures include inserting a tube inside the bowel or oesophagus to open up a blockage; insertion of a 'stent'). Some patients may be advised or may choose not to undergo any form of treatment.

Deciding whether a person is fit enough to undergo a major operation is difficult and depends on patient factors (e.g. heart and lung fitness, other medical conditions, patient choice) and technical factors (location and spread of disease, availability of other options for treatment).

In the outpatient setting there are a number of tests that can be used to try to work out what the risks of a major operation will be for a particular person. These can then guide different approaches to try to lessen these risks. Examples include exercise programmes, dietary supplements and anxiety management programmes in the period before the operation. In the emergency setting there is often not sufficient time before their operation but there are still a number of ways of improving the chances of a good recovery, such as meeting with a physiotherapist and early planning for discharge needs.

This study aims to explore:

1. Whether patients who have poor outcomes after surgery can be identified at the start of their surgical journey
2. Whether there are specific patient characteristics that are associated with whether individual patients undergo major surgery or not.
3. What patients feel about different support measures that may be put in place to try to improve outcomes

DETAILED DESCRIPTION:
The UK population is aging. Under-investigation and under-treatment of older people is common, with rates of surgery declining with age, despite the incidence of surgically treated gastrointestinal pathology increasing with age. There are large variations in outcomes in older people, between different surgical units in the UK, which suggests that not all patients are receiving the same level of care or access to resources. In GI surgery, the concern is that patients in centres with low elective surgery rates will be inappropriately denied the benefits of operative intervention (disease control, symptom improvement), with consequently higher rates of emergency admission and intervention. Conversely, in centres with high rates of elective surgery, patients may be inappropriately subjected to the morbidity or even mortality of surgery with limited or no benefit.

Major surgery remains one of the most debilitating events that an older person may experience and may profoundly influence functional decline and disability. Optimisation of outcomes in older patients with comorbidities and frailty requires multi-professional input which is often lacking. Adverse factors associated with ageing include co-morbidity, polypharmacy, cognitive impairment, dependency and frailty, all of which are associated with increased all cause mortality in the general population. There is also a natural decline in cardiorespiratory fitness with age, however this may be modifiable with physical activity or exercise. Malnutrition and psychological problems are also very common in patients requiring gastrointestinal surgery. When these at-risk individuals are exposed to the stress of major abdominal surgery, post-operative mortality and morbidity also increase. Common lifestyle choices, including smoking, excess alcohol consumption and sedentary behaviours, add to this risk.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 65+ years old inclusive
* Patients with a diagnosis of gastrointestinal pathology amenable to elective, urgent (unscheduled) or emergency major gastrointestinal surgery who either undergo surgery, a risk-adapted procedure or are managed conservatively (due to patient wishes, co-morbidities or frailty).
* Mental capacity to consent

Exclusion Criteria:

* Patients aged less than 65 years old
* Patients with unresectable disease (location, invasion, dissemination)
* Lack mental capacity to consent
* Unable to understand the information provided (translational issues)
* Prisoners
* Patients undergoing surgery for major trauma
* Patients undergoing surgery for primary gynaecological, vascular or urological disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients with GI pathology amenable to surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Functional recovery at 6 weeks post-operation/ definitive procedure or from decision not to operate | 6 weeks
  World Health Organisation Disability Assessment Schedule (WHO DAS). This is scored from 0 to 48 and then converted into a percentage. Minimum score 0%, maximum score 100%. Higher scores denote more disabled. "Disabled" classified as a score of 25% or higher. A change of 8% or more from baseline is defined as a new disability.

SECONDARY OUTCOMES:
Health related quality of life | 6 weeks
  EQ-5D-5L Visual analogue scale (VAS) will be used for statistical analysis which is a scale from 0 to 100 with 0 being the worst health you can imagine and 100 being the best health you can imagine. Baseline score will be compared to post-operative score.
Length of hospital stay | From day 0 (hospital admission) to discharge from hospital (on average 6 days)
  The number of days from hospital admission (day 0) to discharge from hospital (on average 6 days)
Treatment related adverse events | From day 0 (treatment) to discharge from hospital (on average 6 days)
  Reporting the type and grade of adverse event relating to the treatment. The AE will be graded using the Clavien-Dindo Classification system (grades I-IV), grade IV being the most severe.
Survival | 6 months
  Any death 6 months from index procedure or decision

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Daniels, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (2):
- United Kingdom (2):
  - Sheffield Teaching Hospitals NHS FT, Sheffield, Yorkshire
  - Barnsley Hospital NHS FT, Barnsley

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniels SL, Lee MJ, Moug S, Wilson TR, Burton M, George J, Brown SR, Wyld L. Protocol for a multi-centre observational and mixed methods pilot study to identify factors predictive of poor functional recovery after major gastrointestinal surgery and strategies to enhance uptake of perioperative optimization: Optimizing the care and treatment pathways for older patients facing major gastrointestinal surgery (OCTAGON). Colorectal Dis. 2021 Jun;23(6):1552-1561. doi: 10.1111/codi.15603. Epub 2021 Mar 22. PMID 33638249